CLINICAL TRIAL: NCT05055986
Title: Accuracy of Open-source Software in Semi-automatic 3-Dimensional Reconstruction of the Mandible: A Validity and Reliability Study
Brief Title: Accuracy of Open-source Software in Semi-automatic 3-Dimensional Reconstruction of the Mandible
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Sayed Mohamed Shazly, Teaching Assistant, Cairo University
Other Study IDs: Open-source Software
Record Dates: First submitted 2021-09-11; First posted 2021-09-24 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Segmentation; Bone
Keywords: Open source software; Segmentation; Mandible

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CBCT Dicom files of patients: CBCT Dicom files of patients will be used for measurements of mandibular bone volume by open-source software.
  Interventions: Device: Semiautomatic segmentation of open-source software

INTERVENTIONS:
Device: Semiautomatic segmentation of open-source software — Semiautomatic segmentation of open-source software is accurate as of the manual segmentation of commercial software.
  Other Names: ITK-Snap software; 3D Slicer software

SUMMARY:
Concomitant to the evolution of CBCT devices, several post-processing software packages were developed for producing 3D-printed models of anatomical structures. In the last few years, several open-source software used as an alternative to commercial software for 3D reconstruction of anatomical structures such as the mandible. However, no sufficient evidence validating the accuracy of this open-source software.

DETAILED DESCRIPTION:
3D rendering of craniomaxillofacial structures is based on the segmentation process. Semi-automatic segmentation has been pointed out as the technique of choice since it combines the high efficiency and repeatability of the automatic methods with the experience of an operator. Although the creation of 3D models is very important, it is still not a common procedure, since commercial software often requires higher electronic computer power and is licensed by its manufacturer, increasing the financial costs. In the last few years, several open-source software can be obtained for free such as ITK-Snap and 3D Slicer, which could provide more economical options for clinicians or researchers in patient management. However, no sufficient evidence validating the accuracy of this open-source software in detecting the volumetric and morphological characteristics of craniomaxillofacial structures.

ELIGIBILITY:
Inclusion Criteria:

* Good quality CBCT scans.
* Field of view (FOV) including the whole mandibular bone.
* Absence of artifacts, dental implants, craniofacial deformities, and temporomandibular disorders.

Exclusion Criteria:

* Low-quality CBCT scans.
* FOV not including the whole mandibular bone.
* Presence of artifacts, dental implants, craniofacial deformities, and temporomandibular disorders.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who come to the Oral and Maxillofacial Department, Faculty of Dentistry, Cairo University for CBCT imaging for orthodontic treatment. Patients will be with intact mandible and free of any injury or disease that can affect the volume of the mandible.
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Validity and reliability of CBCT open-source software (ITK-Snap and 3D Slicer) semiautomatic segmentation in Volumetric measurement of mandibular bone. | 1 year
  The volume calculation function tool of the dedicated CBCT open-source software (ITK-Snap and 3D Slicer) will be used to measure the mandibular bone volume.

CONTACTS AND LOCATIONS:
Overall Officials: Maha S Mohamed, Master, Principal Investigator — Cairo University
Locations (1):
- Faculty of dentistry cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Gomes AF, Brasil DM, Silva AIV, Freitas DQ, Haiter-Neto F, Groppo FC. Accuracy of ITK-SNAP software for 3D analysis of a non-regular topography structure. Oral Radiol. 2020 Apr;36(2):183-189. doi: 10.1007/s11282-019-00397-y. Epub 2019 Jul 2. PMID 31267257
- [Background] Matsiushevich K, Belvedere C, Leardini A, Durante S. Quantitative comparison of freeware software for bone mesh from DICOM files. J Biomech. 2019 Feb 14;84:247-251. doi: 10.1016/j.jbiomech.2018.12.031. Epub 2018 Dec 21. PMID 30591203
- [Background] Lo Giudice A, Ronsivalle V, Grippaudo C, Lucchese A, Muraglie S, Lagravere MO, Isola G. One Step before 3D Printing-Evaluation of Imaging Software Accuracy for 3-Dimensional Analysis of the Mandible: A Comparative Study Using a Surface-to-Surface Matching Technique. Materials (Basel). 2020 Jun 21;13(12):2798. doi: 10.3390/ma13122798. PMID 32575875
- [Background] Vallaeys K, Kacem A, Legoux H, Le Tenier M, Hamitouche C, Arbab-Chirani R. 3D dento-maxillary osteolytic lesion and active contour segmentation pilot study in CBCT: semi-automatic vs manual methods. Dentomaxillofac Radiol. 2015;44(8):20150079. doi: 10.1259/dmfr.20150079. Epub 2015 May 21. PMID 25996572